CLINICAL TRIAL: NCT03923205
Title: Assessing the Effects of a Buckwheat Beverage on Postprandial Glucose Metabolism on Healthy and T2D Individuals
Acronym: BUCKFOOD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2-088-18
Record Dates: First submitted 2019-04-03; First posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Healthy; Type2 Diabetes
Keywords: buckwheat; postprandial glycemia; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: Three groups ; healthy volunteers, individuals with T2D controlled by medication and individuals with T2D controlled by diet and lifestyle only. All groups follow same interventions assigned randomly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control meal (Active Comparator): The control meal will be a standard OGT test containing 75 g glucose dissolved in 300 mL of water followed by 100 mL water.
  Interventions: Other: Dietary Intervention
- The test meal (Active Comparator): The test meal contains 100 g of the buckwheat beverage and 75 g glucose dissolved in 300 mL water followed by 100 mL water.
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention — The effect of a buckwheat beverage on postprandial glucose metabolism in healthy individuals and those with T2D controlled by medication and diet will be studied.

SUMMARY:
Buckwheat is a unique crop because is naturally rich in compounds that have shown beneficial effects on glucose metabolism.

A constant high glucose level in blood after meal consumption is an independent risk factor for cardiovascular complications and death. In order to prevent Type 2 Diabetes Mellitus (T2D) and/or its complications it is important to have a strict control of the blood glucose levels after a meal. There are known therapies for the control of the high glucose blood levels such as agents that act on intestinal digestion of carbohydrates and therapeutic agents that mimic the insulin response after a meal. The combination of these type of agents was commonly prescribed in the treatment of T2D.

The aim of the study is to assess the effect of a buckwheat beverage on postprandial glucose metabolism in healthy individuals and those with T2D controlled by medication and diet.

DETAILED DESCRIPTION:
The ability of the buckwheat beverage to modulate postprandial sugar metabolism will be tested in a dietary study in healthy volunteers and people with T2D. Three groups will be recruited; healthy volunteers, individuals with T2D controlled by medication and individuals with T2D controlled by diet and lifestyle only.

For the human volunteers who have T2D controlled by medication, there will be targeted those who have been prescribed metformin only.

The volunteers will visit the Human Nutrition Unit (HNU) three times (a screening visit and two study visits) during the course of the study.

A minimum of two weeks between the study visits will be allowed.

Screening visit:

Once the consent form has been signed, the volunteers taking part in the study will answer a specific health questionnaire and have their blood sugar level measured. The HbA1c (glycated haemoglobin) will be measured using the AS-100 (finger spot blood). We will follow the NHS guideline to establish the values for HbA1c. A normal HbA1c target is below 48 mmol/mol (or 6.5%).

In addition, for the volunteers with T2D, a consultant from the study research team will access the medical records to ensure their eligibility for the study. Permission will be obtained from the volunteers for this via the study consent form.

Dietary study test meal and control meal:

The test meal The buckwheat beverage is prepared from sprouted buckwheat flour without adding any extra sugar, spices or aromas. The test meal contains 100 g of the buckwheat beverage and 75 g glucose dissolved in 300 mL water followed by 100 mL water.

The control meal The control meal will be a standard OGT test containing 75 g glucose dissolved in 300 mL of water followed by 100 mL water.

Both meals will be advised to be consumed within 5 minutes. The T2D volunteers which are on metformin will be advised to take their medication as usual. We will record the dose and time when the metformin will be taken by the volunteers.

Dietary study visits:

Following recruitment, screening and consent, the three groups of volunteers will start the study by random allocation to one of the test meals. On the study day, the volunteers will be advised to come to the HNU in the morning after an overnight fasting (10 h). A cannula will be inserted into the volunteers' arm and baseline blood will be collected. The cannulation and blood sampling will be performed by trained phlebotomists. Additionally a baseline urine sample will be collected. The urine sample either will be brought in by the volunteers in the morning or produced in HNU before the test meals. The volunteers will be served the control and test meal (depending on allocation) and advised that it is to be consumed within five minutes. Volunteers which are on metformin will be asked to take their medication as usual.

For each study visit, blood will be collected at 0, 15, 30, 45, 60, 75, 90, 105, 120, 150, 180 and 300 min. The blood will be collected in 4 mL lithium heparin tubes and 4 mL glucose (fluoride oxalate) tubes at each time point. A volume of 96 mL of blood will be collected at each study visit. Additionally a volume of 5 μL blood will be collected for each time point in order to instantly measure the glucose levels. At least two samples will be collected at t=0 in order to obtain a good baseline value.

The movements of the volunteers will be restricted to minimum for the entire blood collection period. They will be asked to stay resting and comfortable position and relaxed for the entire (300 min) sampling period and to not leave the HNU.

After five hours, once all the blood samples have been collected the cannula will be extracted from the volunteer's arm and lunch will be provided.

ELIGIBILITY:
Inclusion Criteria:

Healthy and T2D (controlled by diet and lifestyle or metformin) volunteers; Age 18+; males and females.

Exclusion Criteria:

For the healthy group:

* taking prescribed medication
* HbA1c above 48mmol/mol (or 6.5%)
* pregnant or breastfeeding
* blood donation in the last three months
* unable to give written informed consent
* eating disorders such as anorexia, bulimia, binge eating or night eating syndrome.
* significant health issue
* taking vitamin or mineral supplements (unless they agree to discontinue supplementation 2 weeks or more before the start of the study)
* Food allergies/intolerances

For the T2D groups:

* T2D controlled by medication other than metformin
* pregnant or breastfeeding
* blood donation in the last three months
* unable to give written informed consent
* eating disorders such as anorexia, bulimia, binge eating or night eating syndrome.
* any other significant health issue other than T2D
* taking vitamin or mineral supplements (unless they agree to discontinue supplementation 2 weeks before the start of the study)
* food allergies/intolerances

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2019-03-07 (Actual); Primary Completion 2020-09-07 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
post prandial blood glucose (recording cmax) | five hours
  Postprandial blood glucose levels after acute consumption of a buckwheat beverage, recording the maximum blood glucose concentration (c max) over the baseline after the consumption of a buckwheat beverage.
AUC for postprandial glucose | five hours
  Area under the curve described by the postprandial glucose level during five hours time

SECONDARY OUTCOMES:
post prandial blood insulin in blood ( including AUC) | five hours
  Post prandial blood insulin levels after acute consumption of a buckwheat beverage. AUC (area under curve) for insulin for five hour interval.
Buckwheat beverage key bioactives bioavailability and metabolism. | five hours
  Plasma concentration of key bioactives (inositols and fagomines)
Urine ratio of myo and D-chiro inositol | 0, 3 and 5 hours
  Urine ratio of myo and D-chiro inositol after the consumption of a buckwheat beverage.
Urine glucose concentration | 0, 3 and 5 hours
  Glucose concentration in urine after the consumption of a buckwheat beverage.

CONTACTS AND LOCATIONS:
Locations (1):
- Rowett Institute, University of Aberdeen, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No